CLINICAL TRIAL: NCT03011749
Title: Value of FLT PET/CT in Radium-223 Therapy of Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: Value of FLT PET/CT in Radium-223 Therapy of mCRPC Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marie Øbro Fosbøl, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1603551
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Prostate Carcinoma
Keywords: Radium-223 therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLT PET/CT (Experimental): FLT PET/CT
  Interventions: Other: FLT PET/CT

INTERVENTIONS:
Other: FLT PET/CT — FLT PET/CT before first series of Radium-223 and after 2 series

SUMMARY:
The aim of the study is to investigate whether positron emission tomography (PET) using the tracer 18F-Fluorothymidine (FLT) can provide information on proliferative activity in bone marrow of patients receiving Radium 223 therapy and potentially be a predictive marker of hematological toxicity

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration resistant prostate cancer
* Eligible for Radium-223 therapy
* Informed consent

Exclusion Criteria:

* Inability to understand study protocol
* Extensive metastatic involvement of the axial skeleton ("superscan" on bone scintigraphy)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Uptake of FLT in hematological bone marrow | 3 months

SECONDARY OUTCOMES:
Occurrence of hematological toxicity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark